CLINICAL TRIAL: NCT01303783
Title: A Multicenter, Multifactorial, Randomized, Double-Blind, Placebo-Controlled Dose-Finding Study of Nifedipine GITS and Candesartan in Combination Compared to Monotherapy in Adult Patients With Essential Hypertension
Brief Title: Study of Nifedipine GITS and Candesartan Combination Compared to Monotherapy in Patients With Essential Hypertension
Acronym: DISTINCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14725; 2009-017077-37 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Hypertension, Essential
Keywords: Nifedipine GITS; Candesartan; mild to moderate Hypertension; Combination therapy
MeSH Terms: conditions — Essential Hypertension | interventions — candesartan cilexetil; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (16):
- Nifedipine GITS 20 mg (Experimental): Subjects received 20 mg of nifedipine GITS (single tablet) monotherapy once daily for 8 weeks along with 2 placebo tablets and 1 placebo capsule
  Interventions: Drug: Nifedipine GITS (Adalat, BAYA1040), 20 mg; Drug: Placebo
- Nifedipine GITS 30 mg (Experimental): Subjects received 30 mg of nifedipine GITS (single tablet) monotherapy once daily for 8 weeks along with 2 placebo tablets and 1 placebo capsule
  Interventions: Drug: Nifedipine GITS (Adalat, BAYA1040), 30 mg; Drug: Placebo
- Nifedipine GITS 60 mg (Experimental): Subjects received 60 mg of nifedipine GITS (single tablet) monotherapy once daily for 8 weeks along with 2 placebo tablets and 1 placebo capsule
  Interventions: Drug: Nifedipine GITS (Adalat, BAYA1040), 60 mg; Drug: Placebo
- Candesartan cilexetil 4 mg (Experimental): Subjects received 4 mg of candesartan cilexetil (single capsule) monotherapy once daily for 8 weeks along with 3 placebo tablets
  Interventions: Drug: Candesartan cilexetil (Atacand), 4 mg; Drug: Placebo
- Candesartan cilexetil 8 mg (Experimental): Subjects received 8 mg of candesartan cilexetil (single capsule) monotherapy once daily for 8 weeks along with 3 placebo tablets
  Interventions: Drug: Candesartan cilexetil (Atacand), 8 mg; Drug: Placebo
- Candesartan cilexetil 16 mg (Experimental): Subjects received 16 mg of candesartan cilexetil (single capsule) monotherapy once daily for 8 weeks along with 3 placebo tablets
  Interventions: Drug: Placebo; Drug: Candesartan cilexetil (Atacand), 16 mg
- Candesartan cilexetil 32 mg (Experimental): Subjects received 32 mg of candesartan cilexetil (single capsule) monotherapy once daily for 8 weeks along with 3 placebo tablets
  Interventions: Drug: Placebo; Drug: Candesartan cilexetil (Atacand), 32 mg
- Nifedipine/candesartan 20/4 mg (Experimental): Subjects received the combination of 20 mg of nifedipine GITS/4 mg of candesartan cilexetil once daily for 8 weeks along with 2 placebo tablets
  Interventions: Drug: Candesartan cilexetil (Atacand), 4 mg; Drug: Nifedipine GITS (Adalat, BAYA1040), 20 mg; Drug: Placebo
- Nifedipine/candesartan 20/8 mg (Experimental): Subjects received the combination of 20 mg of nifedipine GITS/8 mg of candesartan cilexetil once daily for 8 weeks along with 2 placebo tablets
  Interventions: Drug: Candesartan cilexetil (Atacand), 8 mg; Drug: Nifedipine GITS (Adalat, BAYA1040), 20 mg; Drug: Placebo
- Nifedipine/candesartan 20/16 mg (Experimental): Subjects received the combination of 20 mg of nifedipine GITS/16 mg of candesartan cilexetil once daily for 8 weeks along with 2 placebo tablets
  Interventions: Drug: Nifedipine GITS (Adalat, BAYA1040), 20 mg; Drug: Placebo; Drug: Candesartan cilexetil (Atacand), 16 mg
- Nifedipine/candesartan 30/8 mg (Experimental): Subjects received the combination of 30 mg of nifedipine GITS/8 mg of candesartan cilexetil once daily for 8 weeks along with 2 placebo tablets
  Interventions: Drug: Candesartan cilexetil (Atacand), 8 mg; Drug: Nifedipine GITS (Adalat, BAYA1040), 30 mg; Drug: Placebo
- Nifedipine/candesartan 30/16 mg (Experimental): Subjects received the combination of 30 mg of nifedipine GITS/16 mg of candesartan cilexetil once daily for 8 weeks along with 2 placebo tablets
  Interventions: Drug: Nifedipine GITS (Adalat, BAYA1040), 30 mg; Drug: Placebo; Drug: Candesartan cilexetil (Atacand), 16 mg
- Nifedipine/candesartan 30/32 mg (Experimental): Subjects received the combination of 30 mg of nifedipine GITS/32 mg of candesartan cilexetil once daily for 8 weeks along with 2 placebo tablets
  Interventions: Drug: Nifedipine GITS (Adalat, BAYA1040), 30 mg; Drug: Placebo; Drug: Candesartan cilexetil (Atacand), 32 mg
- Nifedipine/candesartan 60/16 mg (Experimental): Subjects received the combination of 60 mg of nifedipine GITS/16 mg of candesartan cilexetil once daily for 8 weeks along with 2 placebo tablets
  Interventions: Drug: Nifedipine GITS (Adalat, BAYA1040), 60 mg; Drug: Placebo; Drug: Candesartan cilexetil (Atacand), 16 mg
- Nifedipine/candesartan 60/32 mg (Experimental): Subjects received the combination of 60 mg of nifedipine GITS/32 mg of candesartan cilexetil once daily for 8 weeks along with 2 placebo tablets
  Interventions: Drug: Nifedipine GITS (Adalat, BAYA1040), 60 mg; Drug: Placebo; Drug: Candesartan cilexetil (Atacand), 32 mg
- Placebo (Placebo Comparator): Subjects received placebo (3 tablets and 1 capsule) once daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan cilexetil (Atacand), 4 mg — 4 mg of candesartan as capsule
  Arms: Candesartan cilexetil 4 mg; Nifedipine/candesartan 20/4 mg
Drug: Candesartan cilexetil (Atacand), 8 mg — 8 mg candesartan as capsule
  Arms: Candesartan cilexetil 8 mg; Nifedipine/candesartan 20/8 mg; Nifedipine/candesartan 30/8 mg
Drug: Nifedipine GITS (Adalat, BAYA1040), 20 mg — 20 mg nifedipine as tablet
  Arms: Nifedipine GITS 20 mg; Nifedipine/candesartan 20/16 mg; Nifedipine/candesartan 20/4 mg; Nifedipine/candesartan 20/8 mg
Drug: Nifedipine GITS (Adalat, BAYA1040), 30 mg — 30 mg nifedipine as tablet
  Arms: Nifedipine GITS 30 mg; Nifedipine/candesartan 30/16 mg; Nifedipine/candesartan 30/32 mg; Nifedipine/candesartan 30/8 mg
Drug: Nifedipine GITS (Adalat, BAYA1040), 60 mg — 60 mg nifedipine as tablet
  Arms: Nifedipine GITS 60 mg; Nifedipine/candesartan 60/16 mg; Nifedipine/candesartan 60/32 mg
Drug: Placebo — 3 different placebo tablets corresponding nifedipine doses and 1 placebo capsule corresponding to candesartan doses
Drug: Candesartan cilexetil (Atacand), 16 mg — 16 mg of candesartan as capsule
  Arms: Candesartan cilexetil 16 mg; Nifedipine/candesartan 20/16 mg; Nifedipine/candesartan 30/16 mg; Nifedipine/candesartan 60/16 mg
Drug: Candesartan cilexetil (Atacand), 32 mg — 32 mg of candesartan as capsule
  Arms: Candesartan cilexetil 32 mg; Nifedipine/candesartan 30/32 mg; Nifedipine/candesartan 60/32 mg

SUMMARY:
The purpose of this study is to determine the blood pressure lowering responses of various dose combinations of nifedipine GITS and candesartan as compared to treatment with each component on their own (monotherapy) and placebo (a look-alike tablet without active ingredient). The drugs - nifedipine GITS and candesartan - which are being investigated are currently approved for use in patients with essential hypertension alone or together with other antihypertensive drugs (combination therapy), but the optimal dose of nifedipine GITS and candesartan used together in the treatment of essential hypertension has not been established yet. In this study patients will be treated with various doses of nifedipine GITS and/or candesartan or placebo. These different regimens will be administered once a day and will be assessed based on their blood pressure lowering effects (mean sitting diastolic blood pressure) in subjects with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years or older. Female subjects must be either post-menopausal for one year, surgically sterile, or using an effective contraceptive method. Hormonal contraceptive use is disallowed.
* Subjects must have mild to moderate essential hypertension (Grade 1 and 2 WHO classifications) as measured by calibrated standard sphygmomanometer. (MSDBP of ≥90 mmHg and < 110 mmHg at Visit 1 (placebo run-in), and MSDBP of ≥95 mmHg and < 110 mmHg at visit 2 (randomization)
* Subjects must have an absolute difference in their MSDBP of less than 10 mmHg between Visit 1 (placebo run- in) and Visit 2 (randomization).

Exclusion Criteria:

* Severe hypertension (Grade 3 WHO classification; MSDBP ≥110 mmHg and/or MSSBP ≥ 180 mmHg)
* Inability to washout of antihypertensive drugs (even if prescribed for another indication) safely for a period of 14 weeks.
* History of hypertensive retinopathy - known Keith-Wagener Grade III or IV
* History of hypertensive encephalopathy
* Cerebrovascular ischemic event (stroke, transient ischemic attack [TIA])within the previous 12 months
* History of intracerebral hemorrhage or subarachnoid hemorrhage
* Evidence of secondary hypertension such as coarchation of the aorta, pheochromocytoms, hypersaldosteronism, etc.
* Type I diabetes mellitus (DM) or poorly controlled DM Type II as evidenced by a glycosylated hemoglobin [HbA1C] of greater than 9% on visit 1.
* Allergies or known intolerance to one of the investigational drugs/drug class or to one of their ingredients
* Any history of heart failure, New York Heart Association (NYHA) classification III or IV
* Severe coronary heart disease as manifest by a history of myocardial infarction or unstable angina in the last 6 months prior to visit 1.
* Clinically significant cardiac valvular disease
* History of malignancy in the last 5 years, excluding basal or skin cancer
* Uncorrected hypokalemia or hyperkalemia: potassium outside 3.0-5.0 mmol/L
* Surgical or medical conditions that might alter the metabolism, excretion or distribution or absorption of any drug

  1. Gastrointestinal disease or surgery resulting in the potential for malabsorption
  2. Severe gastrointestinal tract narrowing; kock pouch (ileostomy after proctocolectomy)
  3. Cholestasis or biliary obstruction or history of pancreatic injury or clinical significant increase of lipase, amylase, or bilirubin.
  4. Liver disease or AST/ALT levels >3 x ULN
  5. Renal insufficiency, defined as eGFR of < 50 mL/min (computed using the Cockroft-Gault formula), or on hemodialysis
* Investigation trial participation with receipt of investigational study drug within the last month
* Previous assignment to treatment in this study
* Female subjects who are pregnant or lactating.
* Subjects who have night employment (night shift).
* Subjects with an aortic aneurysm that, in the opinion of the investigator, will be unsuitable to be enrolled in the study.
* Thought by the investigator for any reason to be unsuitable for participation in a clinical study
* Systemic use of known cytochrome P450-3A4 inhibitors (e.g cimetidine, anti-human immunodeficiency virus [HIV] protease inhibitors e.g. ritonavir, azole anti-mycotics eg. ketoconazole,) or inducers (e.g rifampicin, anti-epileptic drugs eg. phenytoin, carbamazepine and phenobarbitone) or some P450-3A4 substrates (e.g quinidine, digoxin, tacrolimus)
* Present severe rhythm or conduction disorder:
* Atrial fibrillation
* Second or third degree heart block without a pacemaker.
* Baseline QTc >450 msec
* History of non-compliance, alcoholism or drug abuse that in the opinion of the investigator will compromise successful completion of the study.
* If differences greater than 20 mmHg for SBP and 10 mmHg for DBP are present on 3 consecutive BP readings, the subject should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1381 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the change from baseline in mean seated diastolic blood pressure (MSDBP) at Week 8 | Baseline taken at Visit 1; primary outcome variable assesed at 8 weeks

SECONDARY OUTCOMES:
Change in mean seated systolic blood pressure (MSSBP) at Week 8 | 8 weeks
Control rate at Week 8 | 8 weeks
Response rate at Week 8 | 8 weeks
Peripheral Edema | 8 weeks
Time to achieve first BP control | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (114):
- United States (21):
  - Mobile, Alabama
  - Los Angeles, California
  - Coral Gables, Florida
  - Deerfield Beach, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Valparaiso, Indiana
  - Charlotte, North Carolina
  - Harrisburg, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Mt. Pleasant, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Kenosha, Wisconsin
- Argentina (8):
  - Bahía Blanca, Buenos Aires
  - Quilmes, Buenos Aires
  - Zárate, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Corrientes, Corrientes Province
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
  - Santa Fe, Santa Fe Province
- Belgium (4):
  - Wetteren, Oost-Vlaanderen
  - De Pinte
  - Deurne
  - Ham
- Brazil (6):
  - Fortaleza, Ceará
  - Brasília, Federal District
  - Goiânia, Goiás
  - Rio de Janeiro, Rio de Janeiro
  - Campinas, São Paulo
  - São Paulo, São Paulo
- Canada (12):
  - Langley, British Columbia
  - St. John's, Newfoundland and Labrador
  - Brampton, Ontario
  - Corunna, Ontario
  - Downsview, Ontario
  - Etobicoke, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Strathroy, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Italy (9):
  - Chieti, Abruzzo
  - Bologna, Emilia-Romagna
  - Trieste, Friuli Venezia Giulia
  - Milan, Lombardy
  - Pavia, Lombardy
  - Sassari, Sardinia
  - Pisa, Tuscany
  - Perugia, Umbria
  - Mercato San Severino
- Lithuania (3):
  - Alytus
  - Kaunas
  - Vilnius
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Smolensk
- South Africa (8):
  - Port Elizabeth, Eastern Cape
  - Johannesburg, Gauteng
  - Petoria, Gauteng
  - Roodepoort, Gauteng
  - Durban, KwaZulu-Natal
  - Witbank, Mpumalanga
  - Somerset West, Western Cape
  - Stellenbosch, Western Cape
- South Korea (9):
  - Daejeon, Daejeon Gwang''yeogsi
  - Wŏnju, Gang''weondo
  - Anyang-si, Gyeonggido
  - Goyang-si, Gyeonggido
  - Uijeongbu-si, Gyeonggido
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Chungchungbuk-do
  - Seoul
- Spain (10):
  - Santiago de Compostela, A Coruña
  - Benidorm, Alicante
  - Petrel, Alicante
  - Barcelona, Barcelona
  - Hostalets de Balenyà, Barcelona
  - Peralada, Girona
  - Granada, Granada
  - Huelva, Huelva
  - Oviedo, Principality of Asturias
  - Valencia, Valencia
- Ukraine (6):
  - Dnipropetrovsk
  - Kharkiv
  - Kiev
  - Vinnitsa
  - Zaporizhzhya
  - Zhytomyr
- United Kingdom (15):
  - Bath, Avon
  - Fowey, Cornwall
  - Penzance, Cornwall
  - St Austell, Cornwall
  - Chesterfield, Derbyshire
  - Glasgow, Glasgow City
  - Blackpool, Lancashire
  - Bath, Somerset
  - Addlestone, Surrey
  - Coventry, Warwickshire
  - Royal Leamington Spa, Warwickshire
  - Chippenham, Wiltshire
  - Trowbridge, Wiltshire
  - Westbury, Wiltshire
  - Bath

REFERENCES:
- [Result] Kjeldsen SE, Cha G, Villa G, Mancia G; DISTINCT Investigators. Nifedipine GITS/Candesartan Combination Therapy Lowers Blood Pressure Across Different Baseline Systolic and Diastolic Blood Pressure Categories: DISTINCT Study Subanalyses. J Clin Pharmacol. 2016 Sep;56(9):1120-9. doi: 10.1002/jcph.712. Epub 2016 Mar 7. PMID 26829251
- [Derived] Kjeldsen SE, Sica D, Haller H, Cha G, Gil-Extremera B, Harvey P, Heyvaert F, Lewin AJ, Villa G, Mancia G; DISTINCT Investigators. Nifedipine plus candesartan combination increases blood pressure control regardless of race and improves the side effect profile: DISTINCT randomized trial results. J Hypertens. 2014 Dec;32(12):2488-98; discussion 2498. doi: 10.1097/HJH.0000000000000331. PMID 25144296
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/